CLINICAL TRIAL: NCT06054763
Title: Traditional Chinese Herbal Medicine Buyang Huanwu Decoction on Visual Acuity and Visual Field in Patients With Normal Tension Glaucoma：a Double-blind, Randomized Controlled Trial
Brief Title: Buyang Huanwu Decoction and Normal Tension Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Liang Hsieh, Physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH112-REC3-126
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Glaucoma; Visual Acuity; Visual Field; Chinese Medicine
MeSH Terms: conditions — Glaucoma | interventions — buyang huanwu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buyang Huanwu Decoction group (Experimental): Oral administration of Buyang Huanwu Decoction (3 grams), two times in a day after breakfast and dinner, for 12 consecutive weeks
  Interventions: Combination Product: Buyang Huanwu Decoction
- Placebo group (Placebo Comparator): the same method as the treatment group, but taking Buyang Huanwu Decoction placebo (90% starch and 10% Buyang Huanwu Decoction)
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Buyang Huanwu Decoction — Buyang Huanwu Decoction is a common prescription for treating stroke. The possible mechanism is to replenish qi, activate blood circulation, and remove blood stasis.
  Arms: Buyang Huanwu Decoction group
Other: Placebo — 90% starch and 10% Buyang Huanwu Decoction
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to test Buyang Huanwu Decoction in normal intra-ocular pressure glaucoma. The main question to answer is: the effect of Buyang Huanwu Decoction and its safety in patients with normal intra-ocular pressure glaucoma.

Participants will take 3 grams of Buyang Huanwu Decoction or placebo for 12 weeks.

Researchers will compare treatment group and placebo group to see if the visual acuity, visual field would be improved.

DETAILED DESCRIPTION:
There is currently no active and effective treatment for normal intra-ocular pressure glaucoma, and glaucoma patients often affect the optic nerve and cause visual acuity and visual field damage. Studies have found that glaucoma patients have less blood flow to the optic nerve, retina and choroid than normal people. Buyang Huanwu Decoction has the functions of invigorating qi, promoting blood circulation and dredging collaterals, and is often used in the treatment of stroke. Therefore, the purpose of this study is to investigate the effect of Buyang Huanwu Decoction on visual acuity, visual field and its safety in patients with normal intra-ocular pressure glaucoma. This study is designed as a randomized, double-blind, controlled clinical trial. A total of 60 subjects with normal intra-ocular pressure glaucoma were randomly divided into: 1) treatment group (30 subjects), oral administration of Buyang Huanwu Decoction (3 grams), two times in a day after breakfast and dinner, for 12 consecutive weeks; 2) control group (30 subjects), the same method as the treatment group, but taking Buyang Huanwu Decoction placebo (90% starch and 10% Buyang Huanwu Decoction). Primary outcome was changes in visual acuity, visual field, and optic nerve fiber layer, and secondary outcome was changes in quality of life scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of normal tension glaucoma for at least 3 months.
* Using less than 1 medicine for glaucoma.
* Without any eye disease other than normal tension glaucoma.
* Writing the Informed Consent Form by themselves.

Exclusion Criteria:

* With other chronic diseases, such as diabetes, hypertension, cancer.
* With polypharmacy.
* Had glaucoma surgery or myopia laser surgery before the study.
* With mental disease and could not finish the study.
* Allergic to Buyang Huanwu Decoction.
* Pregnancy or lactation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in visual acuity | 12 weeks
  The difference of visual acuity between study baseline and the 12 weeks of intervention.